CLINICAL TRIAL: NCT02174601
Title: A Pre-endoscopic Prediction Model for Inadequate Bowel Preparation in Patients Receiving Split Dose Polyethylene Glycol Preparation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2013-0292
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Colonoscopy
Keywords: bowel preparation; coolprep; colonoscopy; prediction model

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- colonoscopy group

SUMMARY:
After written consent for participating in clinical research studies, all clinical studies conducted to in the one day. The investigators will ask and record about bowel cleansing state in all patients who performed colonoscopy. There is no additional cost and the expected complications.

Based on answer, the investigators will develop a prediction model for inadequate bowel preparation and prove validation. This model can take the additional measures to subjects predicting improper cleansing. It can contribute to improve the accuracy of the test and reduce the discomfort due to re-performing colonoscopy after re-preparation, as well as cost savings due to reduced frequency of re-colonoscopy Ultimately, it will be able to bring a improvement of the quality of management

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old

Exclusion Criteria:

* Less than 20 years old
* Cardiac, renal, and metabolic dysfunction in patients with serious adverse
* Mental or central nervous system disorders
* Individuals with bwel obstruction
* Individuals who can not read and understand the consent form (literacy, foreign, etc.) However, although individuals with vision / hearing disturbance and deterioration of cognitive abilities, they may participate in the research if can be able to complete the survey with one guardian or the help of researchers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects, more than 20 years old, who admitted to the health promotion center for performing colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
bowel cleansing state | average 24hours before colonoscopy after taking coolprep
  Based on quality of bowel preparation(bowel cleansing state), we will develop a prediction model for inadequate bowel preparation. And then, assess to efficiency and reducing subjects' satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance hospital, Seoul, Seoul, South Korea